CLINICAL TRIAL: NCT01581502
Title: Stroke Acute Management With Urgent Risk-factor Assessment and Improvement (SAMURAI) Study on Anticoagulant Therapy in Nonvalvular Atrial Fibrillation (NVAF)
Brief Title: SAMURAI-NVAF Study: Anticoagulant Therapy for Japanese Stroke Patients With Nonvalvular Atrial Fibrillation (NVAF)
Acronym: SAMURAI-NVAF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Principal Investigator, Kazunori Toyoda, National Cerebral and Cardiovascular Center, Ministry of Health, Labour and Welfare, Japan
Other Study IDs: samurai2011; samurai nvaf 2011 (Registry Identifier: SAMURAI study investigators)
Record Dates: First submitted 2012-04-16; First posted 2012-04-20 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Stroke, Acute; Atrial Fibrillation
Keywords: Anticoagulation; Recurrent stroke; Bleeding
MeSH Terms: conditions — Stroke; Atrial Fibrillation; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NVAF, acute ischemic stroke/TIA: Consecutive acute ischemic stroke/TIA patients with nonvalvular atrial fibrillation; most of these patients begin to receive anticoagulant therapy after index stroke/TIA for secondary prevention
  Interventions: Other: This is an observational study.

INTERVENTIONS:
Other: This is an observational study. — This is an observational, not intervention, study.

SUMMARY:
The purpose of this study is to determine choice of anticoagulant therapy during acute and chronic stages of ischemic stroke/TIA and short- and long-term outcomes, including stroke recurrence and bleeding complications, in patients having nonvalvular atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive acute ischemic stroke/TIA patients with NVAF

Exclusion Criteria:

1. Rheumatic mitral valve disease
2. A history of prosthetic valve replacement or mitral valve surgical repair
3. Active infective endocarditis
4. Patient, family member or legally responsible person does not have given informed consent
5. Inappropriate patient's conditions for study enrollment in the opinion of the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: inpatients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Ischemic events | 2 years
  Recurrence of ischemic stroke/TIA, ACS, systemic embolism, aortic dissection, rupture of aortic aneurysm, peripheral artery disease (required hospitalization), VTE, revascularization (including CEA/CAS, PCI, etc)
major bleeding | 2 years
  Major bleeding according to the ISTH definition, including fatal bleeding, intracranial hemorrhage, etc

SECONDARY OUTCOMES:
modified Rankin Scale | 2 years
  modified Rankin Scale
Modification of anticoagulant medication | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kazunori Toyoda, MD, Principal Investigator — SAMURAI Study Investigators
Locations (16):
- Japan (16):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Toyota Memorial Hospital, Toyota, Aichi-ken
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Brain Attack Center Ota Memorial Hospital, Fukuyama, Hiroshima
  - Nakamura Memorial Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - National Hospital Organization Kagoshima Medical Center, Kagoshima, Kagoshima-ken
  - St Marianna University School of Medicine, Kawasaki, Kanagawa
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto, Kyoto
  - South Miyagi Medical Center, Ōkawara, Miyagi
  - Kohnan Hospital, Sendai, Miyagi
  - Kawasaki Medical School, Kurashiki, Okayama-ken
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Jichi Medical University School of Medicine, Shimotsuke, Tochigi
  - Kyorin University School of Medicine, Mitaka, Tokyo

REFERENCES:
- [Result] Toyoda K, Arihiro S, Todo K, Yamagami H, Kimura K, Furui E, Terasaki T, Shiokawa Y, Kamiyama K, Takizawa S, Okuda S, Okada Y, Kameda T, Nagakane Y, Hasegawa Y, Mochizuki H, Ito Y, Nakashima T, Takamatsu K, Nishiyama K, Kario K, Sato S, Koga M; SAMURAI Study Investigators. Trends in oral anticoagulant choice for acute stroke patients with nonvalvular atrial fibrillation in Japan: the SAMURAI-NVAF study. Int J Stroke. 2015 Aug;10(6):836-42. doi: 10.1111/ijs.12452. Epub 2015 Jan 12. PMID 25581108
- [Result] Toyoda K. Is anticoagulant therapy unnecessary for lower-risk Japanese patients with atrial fibrillation? Lessons from the SAMURAI-NVAF and BAT studies. Circ J. 2015;79(2):307-9. doi: 10.1253/circj.CJ-14-1350. Epub 2014 Dec 24. No abstract available. PMID 25744752
- [Derived] Tanaka K, Miwa K, Takagi M, Sasaki M, Yakushiji Y, Kudo K, Shiozawa M, Tanaka J, Nishihara M, Yamaguchi Y, Fujita K, Honda Y, Kawano H, Ide T, Yoshimura S, Koga M, Hirano T, Toyoda K. Increased Cerebral Small Vessel Disease Burden With Renal Dysfunction and Albuminuria in Patients Taking Antithrombotic Agents: The Bleeding With Antithrombotic Therapy 2. J Am Heart Assoc. 2022 Mar 15;11(6):e024749. doi: 10.1161/JAHA.121.024749. Epub 2022 Mar 5. PMID 35253443
- [Derived] Tanaka K, Koga M, Lee KJ, Kim BJ, Mizoguchi T, Park EL, Lee J, Yoshimura S, Cha JK, Lee BC, Koge J, Bae HJ, Toyoda K; CRCS-K Investigators, the SAMURAI Study Investigators. Transesophageal Echocardiography in Ischemic Stroke With Atrial Fibrillation. J Am Heart Assoc. 2021 Nov 16;10(22):e022242. doi: 10.1161/JAHA.121.022242. Epub 2021 Nov 6. PMID 34743551
- [Derived] Tanaka K, Koga M, Lee KJ, Kim BJ, Park EL, Lee J, Mizoguchi T, Yoshimura S, Cha JK, Lee BC, Nakahara J, Suzuki N, Bae HJ, Toyoda K; CRCS-K Investigators and the SAMURAI Study Investigators. Atrial Fibrillation-Associated Ischemic Stroke Patients With Prior Anticoagulation Have Higher Risk for Recurrent Stroke. Stroke. 2020 Apr;51(4):1150-1157. doi: 10.1161/STROKEAHA.119.027275. Epub 2020 Feb 26. PMID 32098607
- [Derived] Mizoguchi T, Tanaka K, Toyoda K, Yoshimura S, Itabashi R, Takagi M, Todo K, Shiozawa M, Yagita Y, Yoshimoto T, Terasaki T, Yamagami H, Takizawa S, Inoue M, Kamiyama K, Ihara M, Okada Y, Kitazono T, Koga M; SAMURAI Study Investigators. Early Initiation of Direct Oral Anticoagulants After Onset of Stroke and Short- and Long-Term Outcomes of Patients With Nonvalvular Atrial Fibrillation. Stroke. 2020 Mar;51(3):883-891. doi: 10.1161/STROKEAHA.119.028118. Epub 2020 Jan 22. PMID 31964290
- [Derived] Tokunaga K, Koga M, Itabashi R, Yamagami H, Todo K, Yoshimura S, Kimura K, Sato S, Terasaki T, Inoue M, Shiokawa Y, Takagi M, Kamiyama K, Tanaka K, Takizawa S, Shiozawa M, Okuda S, Okada Y, Kameda T, Nagakane Y, Hasegawa Y, Shibuya S, Ito Y, Matsuoka H, Takamatsu K, Nishiyama K, Kario K, Yagita Y, Fujita K, Ando D, Kumamoto M, Arihiro S, Toyoda K; SAMURAI Study Investigators. Prior Anticoagulation and Short- or Long-Term Clinical Outcomes in Ischemic Stroke or Transient Ischemic Attack Patients With Nonvalvular Atrial Fibrillation. J Am Heart Assoc. 2019 Feb 5;8(3):e010593. doi: 10.1161/JAHA.118.010593. PMID 30691339
- [Derived] Koga M, Yoshimura S, Hasegawa Y, Shibuya S, Ito Y, Matsuoka H, Takamatsu K, Nishiyama K, Todo K, Kimura K, Furui E, Terasaki T, Shiokawa Y, Kamiyama K, Takizawa S, Okuda S, Okada Y, Kameda T, Nagakane Y, Yagita Y, Kario K, Shiozawa M, Sato S, Yamagami H, Arihiro S, Toyoda K; SAMURAI Study Investigators. Higher Risk of Ischemic Events in Secondary Prevention for Patients With Persistent Than Those With Paroxysmal Atrial Fibrillation. Stroke. 2016 Oct;47(10):2582-8. doi: 10.1161/STROKEAHA.116.013746. Epub 2016 Aug 16. PMID 27531346